CLINICAL TRIAL: NCT05611957
Title: A Parallel-group, Phase 1, Open-label Study to Investigate the Pharmacokinetics of LY3437943 in Participants With Renal Impairment Compared With Healthy Participants
Brief Title: A Study of LY3437943 in Healthy Participants and Participants With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18529; J1I-MC-GZBL (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09-15

CONDITIONS: Healthy; Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — retatrutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3437943 (Control) (Experimental): LY3437943 administered subcutaneous (SC) to participants with normal renal function
  Interventions: Drug: LY3437943
- LY3437943 (Severe Renal Impairment) (Experimental): LY3437943 administered SC to participants with severe renal impairment
  Interventions: Drug: LY3437943
- LY3437943 (End-Stage Renal Disease) (Experimental): LY3437943 administered SC to participants with end-stage renal disease
  Interventions: Drug: LY3437943

INTERVENTIONS:
Drug: LY3437943 — Administered SC.

SUMMARY:
The main purpose of this study is to assess the amount of study drug that reaches the bloodstream and the time it takes for the body to get rid of it when given to participants with renal (kidney) impairment compared to healthy participants. The study will last up to 5 weeks, excluding screening.

ELIGIBILITY:
Inclusion Criteria:

Normal Participants:

* Healthy male and female participants as determined by physical examination
* Participants with normal renal function assessed by estimated glomerular filtration rate (eGFR) ≥ 90 milliliter per minute (mL/min).
* Body mass index (BMI) ≥ 19.0 and ≤ 40.0 kilograms per meter squared (kg/m²)
* Male participants who agree to use contraception and female participants of child bearing potential must agree to use contraceptive methods and women not of child bearing potential can participate.

Participants with Renal Impairment:

* Have acceptable blood pressure (BP) and pulse rate, as determined by the investigator
* Participants with type 2 diabetes must have a glycated hemoglobin (HbA1c) ≥ 5.0% and ≤ 11.5%
* Are males or females with severe renal impairment as determined by a stable eGFR <30 mL/min, not requiring hemodialysis OR
* Are males or females with end-stage renal disease (have received hemodialysis for at least 3 months)

Exclusion Criteria:

* Have known allergies to LY3437943 or related compounds
* Have a current, functioning organ transplant. Nonfunctional renal allografts may be allowed
* Have any abnormality in the 12-lead electrocardiogram (ECG)
* Are women with a positive pregnancy test or women who are lactating

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area under the concentration versus time curve from time zero to infinity (AUC0-∞) of LY3437943 | Predose up to 31 days postdose
  PK: AUC0-∞ of LY3437943
PK: Maximum observed concentration (Cmax) of LY3437943 | Predose up to 31 days postdose
  PK: Cmax of LY3437943

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Orange County Research Center, Tustin, California
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Nucleus Networks, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No